CLINICAL TRIAL: NCT00627926
Title: A Phase 3 Study of 2 Dose Regimens of Telaprevir in Combination With Peginterferon Alfa-2a (Pegasys®) and Ribavirin (Copegus®) in Treatment-Naive Subjects With Genotype 1 Chronic Hepatitis C
Brief Title: A Phase 3 Study of Telaprevir in Combination With Pegasys® and Copegus® in Treatment-Naive Subjects With Genotype 1 Hepatitis C Virus (HCV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX07-950-108
Record Dates: First submitted 2008-02-22; First posted 2008-03-04 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Hepatitis C
Keywords: Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; telaprevir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week (Placebo Comparator): Placebo (PBO) matched to telaprevir 750 mg tablet thrice daily for 12 weeks in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (RBV) tablet orally twice daily at a dose of 1000 milligram per day (mg/day) for subjects weighing less than (<) 75 kilogram (kg) and 1200 mg/day for subjects weighing greater than or equal to (>=) 75 kg, for 48 weeks.
  Interventions: Biological: Pegylated Interferon Alfa 2a; Drug: Ribavirin; Other: Placebo
- Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week (Experimental): Telaprevir 750 mg tablet thrice daily for 8 weeks, then PBO matched to Telaprevir 750 mg tablet thrice daily for 4 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 24 to 48 weeks depending on individual response to telaprevir treatment.
  Interventions: Biological: Pegylated Interferon Alfa 2a; Drug: Telaprevir; Drug: Ribavirin; Other: Placebo
- Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week (Experimental): Telaprevir 750 mg tablet thrice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing >=75 kg, for 24 to 48 weeks depending on individual response to telaprevir treatment.
  Interventions: Biological: Pegylated Interferon Alfa 2a; Drug: Telaprevir; Drug: Ribavirin

INTERVENTIONS:
Biological: Pegylated Interferon Alfa 2a — subcutaneous injection, 180 micrograms once per week
  Other Names: Pegasys, Peg-IFN-alfa-2a
Drug: Telaprevir — 375 mg tablets administered orally every 8 hours at a dose of 750 mg
  Other Names: VX-950
  Arms: Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Drug: Ribavirin — 200 mg tablets administered orally twice daily at a dose of 1000 mg/day for subjects weighing <75 kg and 1200 mg/day for subjects weighing ≥75 kg
  Other Names: Copegus, RBV
Other: Placebo — Telaprevir matching placebo
  Arms: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week; Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week

SUMMARY:
A Phase 3 study to evaluate the efficacy and safety of two dosing regimens of telaprevir in combination with pegylated interferon alfa 2a (Peg-IFN-alfa-2a) and ribavirin (RBV).

ELIGIBILITY:
Inclusion Criteria

* Has not received any previous treatment with any approved or investigational drug or drug regimen for the treatment of hepatitis C
* Male and female subjects, 18 to 70 years of age, inclusive
* Genotype 1, chronic hepatitis C with detectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
* Screening laboratory values, tests, and physical exam within acceptable ranges
* Able and willing to follow contraception requirements
* Able to read and understand, and willing to sign the informed consent form and abide by the study restrictions

Exclusion Criteria

* Subject has any contraindications to Pegasys® or Copegus® therapy
* Evidence of hepatic decompensation in cirrhotic subjects
* History of organ transplant
* History of, or any current medical condition which could impact the safety of the subject in participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1095 (Actual)
Dates: Start 2008-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (102):
- United States (51):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Fresno, California
  - La Jolla, California
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Carmel, Indiana
  - Indianapolis, Indiana
  - Portland, Maine
  - Baltimore, Maryland
  - Laurel, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Manhasset, New York
  - New York, New York
  - Valhalla, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Annandale, Virginia
  - Charlottesville, Virginia
  - Richmond, Virginia
- Buenos Aires, Argentina
- Australia (7):
  - Darlinghurst
  - Fitzroy
  - Greenslopes
  - Melbourne
  - Perth
  - Westmead
  - Woolloongabba
- Austria (2):
  - Linz
  - Vienna
- Canada (4):
  - Calgary
  - Toronto
  - Vancouver
  - Winnipeg
- France (8):
  - Clichy
  - Créteil
  - Grenoble
  - Lyon
  - Nice
  - Paris
  - Pessac
  - Toulouse
- Germany (9):
  - Berlin
  - Bochum
  - Cologne
  - Düsseldorf
  - Frankfurt
  - Freiburg im Breisgau
  - Hamburg
  - Hanover
  - München
- Israel (5):
  - Haifa
  - Jerusalem
  - Nazareth
  - Petah Tikva
  - Tel Litwinsky
- Italy (3):
  - Bologna
  - Milan
  - Torino
- Poland (6):
  - Bialystok
  - Czeladź
  - Kielce
  - Krakow
  - Lodz
  - Wroclaw
- Santurce, Puerto Rico
- Spain (2):
  - Barcelona
  - Valencia
- United Kingdom (3):
  - Glasgow
  - Hampstead
  - London

REFERENCES:
- [Derived] Jacobson IM, McHutchison JG, Dusheiko G, Di Bisceglie AM, Reddy KR, Bzowej NH, Marcellin P, Muir AJ, Ferenci P, Flisiak R, George J, Rizzetto M, Shouval D, Sola R, Terg RA, Yoshida EM, Adda N, Bengtsson L, Sankoh AJ, Kieffer TL, George S, Kauffman RS, Zeuzem S; ADVANCE Study Team. Telaprevir for previously untreated chronic hepatitis C virus infection. N Engl J Med. 2011 Jun 23;364(25):2405-16. doi: 10.1056/NEJMoa1012912. PMID 21696307

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1095 subjects were enrolled, of which 7 subjects discontinued the study prior to study drug administration. A total of 1088 subjects started treatment.
Period: Overall Study
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Started | 361 | 364 | 363
Completed | 202 | 260 | 268
Not Completed | 159 | 104 | 95
Not completed — Adverse Event | 26 | 37 | 36
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 3 | 4
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Lack of Efficacy | 118 | 40 | 38
Not completed — Noncompliance/unspecified | 8 | 23 | 17

BASELINE CHARACTERISTICS:
Population: The full analysis (FA) set included all randomized subjects who received at least 1 dose of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Total
Number analyzed (Participants) | 361 | 364 | 363 | 1088
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 357 | 359 | 353 | 1069
  >=65 years | 3 | 5 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (10.0) | 47.0 (10.9) | 46.5 (10.8) | 46.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 153 | 149 | 452
  Male | 211 | 211 | 214 | 636
Region of Enrollment [Number; unit: participants]
  North America | 214 | 227 | 214 | 655
  Europe | 106 | 100 | 104 | 310
  Argentina | 8 | 6 | 3 | 17
  Australia | 14 | 14 | 18 | 46
  Israel | 19 | 17 | 24 | 60

OUTCOME MEASURES:

1. Secondary Outcome: Number of Subjects With Undetectable HCV RNA at Week 72
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL and the lower limit of detection was 10 IU/mL.
Time Frame: Week 72 (24 weeks after last dose for subjects with a planned treatment duration of 48 weeks and 48 weeks after last dose for subjects with planned treatment duration of 24 weeks)
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants | 158 | 243 | 265
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 23.0, 95% CI 2-sided [15.9 to 30.0]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 29.2, 95% CI 2-sided [22.4 to 36.1]

2. Secondary Outcome: Number of Subjects Achieving Rapid Viral Response (RVR), Demonstrated by Achieving Undetectable HCV RNA 4 Weeks After Starting Study Treatment
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL and the lower limit of detection was 10 IU/mL. RVR was defined as undetectable HCV RNA 4 weeks after the start of study treatment.
Time Frame: Week 4
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants | 34 | 242 | 246
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 57.1, 95% CI 2-sided [51.4 to 62.8]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 58.4, 95% CI 2-sided [52.7 to 64.0]

3. Secondary Outcome: Number of Subjects Achieving Extended Rapid Viral Response (eRVR), Demonstrated by Achieving Undetectable HCV RNA at Week 4 and at Week 12
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL and the lower limit of detection was 10 IU/mL. eRVR was defined as undetectable HCV RNA at both Week 4 and Week 12.
Time Frame: Week 4 and Week 12
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants | 29 | 207 | 212
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 48.8, 95% CI 2-sided [43.0 to 54.6]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 50.4, 95% CI 2-sided [44.6 to 56.2]

4. Secondary Outcome: Number of Subjects With Undetectable HCV RNA at Week 12
Description: as for outcome 1
Time Frame: Week 12
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants | 146 | 277 | 283
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 35.7, 95% CI 2-sided [29.0 to 42.4]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 37.5, 95% CI 2-sided [30.9 to 44.1]

5. Secondary Outcome: Number of Subjects With Undetectable HCV RNA at End of Treatment (EOT)
Description: as for outcome 1
Time Frame: End of treatment (up to Week 48)
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants | 229 | 295 | 314
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 17.6, 95% CI 2-sided [11.2 to 24.0]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 23.1, 95% CI 2-sided [17.0 to 29.2]

6. Secondary Outcome: Number of Subjects With Undetectable HCV RNA 12 Weeks After Last Planned Dose of Study Treatment
Description: as for outcome 1
Time Frame: 12 weeks after last planned dose of study treatment (up to Week 60)
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants | 161 | 255 | 275
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 25.5, 95% CI 2-sided [18.5 to 32.4]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 31.2, 95% CI 2-sided [24.4 to 37.9]

7. Secondary Outcome: Number of Subjects With Undetectable HCV RNA 24 Weeks After Last Actual Dose of Study Treatment
Description: as for outcome 1
Time Frame: 24 weeks after last actual dose of study treatment (up to Week 72)
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants | 158 | 251 | 274
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 25.2, 95% CI 2-sided [18.2 to 32.2]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; Test type: Superiority or Other; Difference in percentage = 31.7, 95% CI 2-sided [24.9 to 38.5]

8. Secondary Outcome: Number of Subjects With Viral Relapse Planned and Viral Relapse Actual
Description: Viral relapse was defined as having detectable HCV RNA during antiviral follow-up. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL and the lower limit of detection was 10 IU/mL. For viral relapse, 2 analyses were performed: planned and actual. The planned analyses was measured from the end of treatment (EOT) visit to 24 weeks after the last planned dose of study treatment. The actual analyses was measured from the EOT visit to 24 weeks after the last actual dose of study treatment.
Time Frame: After last dose of study drug up to 24 week antiviral follow-up (up to Week 72)
Population: Analysis population included subjects who completed their assigned study drug treatment and had undetectable HCV RNA at the completion of treatment (up to Week 48).
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 229 | 295 | 314
participants
  Viral Relapse Planned | 64 | 28 | 27
  Viral Relapse Actual | 64 | 28 | 25

9. Secondary Outcome: Biochemical Response: Number of Subjects With Grade 3 and 4 Shifts From Baseline in Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) Levels
Description: Criteria for grading severity (toxicity) of ALT and AST: Grade 0 (<1.25*upper limit of normal [ULN]); Grade 1 (mild=1.25 to 2.5*ULN); Grade 2 (moderate=2.6 to 5.0*ULN); Grade 3 (severe= greater than 5.0 to 20.0*ULN); Grade 4 (life-threatening= greater than 20.0*ULN). Number of subjects with Grade 3 shift (from Grade 0, Grade 1 or Grade 2 baseline) and Grade 4 shift (from Grade 0, Grade 1, Grade 2 or Grade 3 baseline) are reported. If a subject experienced more than 1 severity grade shifts during post baseline assessments, the maximum severity grade shift was considered.
Time Frame: Baseline up to Week 48
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants
  ALT Grade 3 toxicity grade shift | 12 | 5 | 6
  ALT Grade 4 toxicity grade shift | 0 | 1 | 0
  AST Grade 3 toxicity grade shift | 19 | 7 | 10
  AST Grade 4 toxicity grade shift | 1 | 0 | 0

10. Secondary Outcome: Noninvasive Markers of Fibrosis: Number of Subjects With Improvement in FibroTest Analysis
Description: FibroTest analysis was a biomarker analysis test used to generate a score that was correlated with the degree of liver damage. The FibroTest score was calculated from the results of a six-parameter blood test, combining six serum markers (alpha-2-macroglobulin, haptoglobin, apolipoprotein A1, gamma-glutamyl transpeptidase, total bilirubin, and alanine transaminase). The FibroTest score (F score) may range from 0.00 (Grade F0) to 1.00 (Grade F4), where F0= no fibrosis and F4=cirrhosis. Results were presented separately for subjects who achieved SVR at 24 weeks after the last planned dose of study treatment and those who did not achieve SVR at 24 weeks after the last planned dose of study treatment. Improvement was defined as decrease of at least 1 grade relative to baseline.
Time Frame: Baseline through 24 weeks after last planned dose of study treatment (up to Week 72)
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug. Here "number of participants analyzed" signifies those subjects who were evaluable for FibroTest Analysis and "n" signifies those subjects who were evaluable for FibroTest Analysis in specified category for each treatment arm, respectively.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 273 | 233 | 261
participants
  SVR achieved (136, 180, 214) | 35 | 59 | 84
  SVR not achieved (137, 53, 47) | 31 | 12 | 12

11. Secondary Outcome: Fatigue Severity Scale (FSS) Total Score
Description: FSS was a 9-item questionnaire where each item was scored on a scale of 1 to 7 (higher scores indicated higher influence of fatigue). FSS total score was calculated as the average of individual items on the questionnaire and FSS total score ranged from 1 to 7, where higher score indicated higher influence of fatigue.
Time Frame: Baseline, Week 4, 12, 24, 36, 48, 72
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug. Here "n" signifies those participants who were evaluable for this measure at given time points for each group, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
units on a scale
  Baseline (n=343, 351, 346) | 3.0 (1.66) | 3.2 (1.63) | 3.0 (1.72)
  Week 4 (n=334, 326, 329) | 4.1 (1.74) | 4.4 (1.74) | 4.5 (1.75)
  Week 12 (n=329, 310, 312) | 4.4 (1.69) | 4.4 (1.68) | 4.8 (1.68)
  Week 24 (n=317, 307, 304) | 4.3 (1.73) | 4.3 (1.71) | 4.3 (1.79)
  Week 36 (n=296, 282, 297) | 4.1 (1.80) | 3.4 (1.84) | 3.3 (1.86)
  Week 48 (n=286, 282, 294) | 4.0 (1.82) | 3.0 (1.75) | 3.1 (1.85)
  Week 72 (n=296, 270, 289) | 2.9 (1.77) | 2.6 (1.56) | 2.6 (1.67)

12. Primary Outcome: Number of Subjects Achieving Sustained Viral Response (SVR), Demonstrated by Achieving Undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels 24 Weeks After Last Planned Dose of Study Treatment
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 international units per milliliter (IU/mL) and the lower limit of detection was 10 IU/mL. Two results are reported: 1) Protocol defined SVR: undetectable HCV RNA at 24 weeks after the last planned dose of study treatment without any confirmed detectable HCV RNA between end of treatment visit (up to Week 48) and 24 weeks after last planned dose (up to Week 72); 2) SVR as per FDA guidance (snapshot analysis): undetectable HCV RNA at 24 weeks after the last planned dose of study treatment. Analysis was based only on the HCV RNA assessment in visit window (+/-2 weeks); if there were more than 1 assessment in the window, the last measurement was used.
Time Frame: 24 weeks after last planned dose of study treatment (up to Week 72)
Population: The full analysis (FA) set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants
  SVR: Protocol Defined | 158 | 250 | 271
  SVR: FDA Guidance | 166 | 261 | 285
Statistical Analysis 1: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; SVR Protocol Defined: undetectable HCV RNA at 24 weeks after the last planned dose of study treatment without any confirmed detectable HCV RNA between end of treatment visit (up to Week 48) and 24 weeks after last planned dose (up to Week 72); Test type: Superiority or Other; Difference in percentage = 24.9, 95% CI 2-sided [17.9 to 31.9]
Statistical Analysis 2: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; Difference in percentage = 30.9, 95% CI 2-sided [24.1 to 37.7]
Statistical Analysis 3: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; SVR FDA Guidance: undetectable HCV RNA at 24 weeks after the last planned dose of study treatment. Analysis was based only on the HCV RNA assessment in visit window (+/-2 weeks); if there were more than 1 assessment in the window, the last measurement was used; Test type: Superiority or Other; Difference in percentage = 25.7, 95% CI 2-sided [18.8 to 32.6]
Statistical Analysis 4: Comparison: PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week vs Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week; [analysis description as in outcome 12, analysis 3]; Test type: Superiority or Other; Difference in percentage = 32.5, 95% CI 2-sided [25.9 to 39.2]

13. Secondary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any adverse change from the subject's baseline (pre-treatment) condition, including any adverse experience, abnormal recording or clinical laboratory assessment value which occurs during the course of the study, whether it is considered related to the study drug or not. An adverse event includes any newly occurring event or previous condition that has increased in severity or frequency since the administration of study drug. SAE: medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event. "Study drug" includes all investigational agents (including placebo, if applicable) administered during the course of the study.
Time Frame: Baseline up to Week 48
Population: The FA set included all randomized subjects who received at least 1 dose of any study drug.
Measure: Number; unit: participants
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Number analyzed (Participants) | 361 | 364 | 363
participants
  AEs | 354 | 362 | 361
  SAEs | 24 | 31 | 33

ADVERSE EVENTS:
Time Frame: AEs and SAEs During Dosing From Baseline to Week 48
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week
Serious Adverse Events (participants affected / at risk) | 24/361 | 31/364 | 33/363
Other Adverse Events (participants affected / at risk) | 354/361 | 362/364 | 361/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week (N=361) | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week (N=364) | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week (N=363)
Cellulitis (Infections and infestations) | 1 | 1 | 1
pneumonia (Infections and infestations) | 0 | 2 | 1
appendicitis (Infections and infestations) | 1 | 0 | 1
lobar pneumonia (Infections and infestations) | 0 | 1 | 1
pyelonephritis (Infections and infestations) | 1 | 1 | 0
urinary tract infection (Infections and infestations) | 0 | 0 | 2
abscess (Infections and infestations) | 0 | 0 | 1
abscess limb (Infections and infestations) | 0 | 1 | 0
acute sinusitis (Infections and infestations) | 0 | 1 | 0
bacteraemia (Infections and infestations) | 0 | 0 | 1
cellulitis staphylococcal (Infections and infestations) | 0 | 1 | 0
escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0
gastroenteritis (Infections and infestations) | 0 | 1 | 0
gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
lung abscess (Infections and infestations) | 0 | 1 | 0
lymphangitis (Infections and infestations) | 0 | 1 | 0
perirectal abscess (Infections and infestations) | 1 | 0 | 0
respiratory tract infection (Infections and infestations) | 0 | 0 | 1
staphylococcal abscess (Infections and infestations) | 0 | 0 | 1
staphylococcal infection (Infections and infestations) | 0 | 0 | 1
subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
tuberculosis (Infections and infestations) | 1 | 0 | 0
anemia (Blood and lymphatic system disorders) | 4 | 10 | 8
neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
anemia haemolytic (Blood and lymphatic system disorders) | 0 | 1 | 0
leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
anal fistula (Gastrointestinal disorders) | 1 | 0 | 0
colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0
inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
internal hernia (Gastrointestinal disorders) | 0 | 1 | 0
intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
salivary gland calculus (Gastrointestinal disorders) | 0 | 1 | 0
syncope (Nervous system disorders) | 0 | 0 | 3
convulsion (Nervous system disorders) | 2 | 0 | 0
migraine (Nervous system disorders) | 1 | 1 | 0
altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
global amnesia (Nervous system disorders) | 1 | 0 | 0
anxiety (Psychiatric disorders) | 1 | 0 | 1
completed suicide (Psychiatric disorders) | 1 | 0 | 0
depression (Psychiatric disorders) | 0 | 1 | 0
insomnia (Psychiatric disorders) | 1 | 0 | 0
panic attack (Psychiatric disorders) | 1 | 0 | 0
psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
intervertebral disc (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
atrial fibrillation (Cardiac disorders) | 1 | 0 | 1
angina pectoris (Cardiac disorders) | 1 | 0 | 0
palpitations (Cardiac disorders) | 1 | 0 | 0
renal failure acute (Renal and urinary disorders) | 2 | 0 | 0
nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
urinary retention (Renal and urinary disorders) | 1 | 0 | 0
retinal exudates (Eye disorders) | 0 | 1 | 0
retinal haemorrhage (Eye disorders) | 0 | 0 | 1
vision blurred (Eye disorders) | 1 | 0 | 0
cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1
hypotension (Vascular disorders) | 0 | 1 | 0
phlebitis (Vascular disorders) | 0 | 0 | 1
thrombophlebitis (Vascular disorders) | 1 | 0 | 0
chest pain (General disorders) | 0 | 0 | 1
non-cardiac chest pain (General disorders) | 0 | 0 | 1
dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
urachal abnormality (Congenital, familial and genetic disorders) | 0 | 0 | 1
cryoglobulinaemia (Immune system disorders) | 1 | 0 | 0
thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PBO 12 Week+Peg-IFN-alfa-2a, RBV 48 Week (N=361) | Telaprevir 8 Week, PBO 4 Week+Peg-IFN-alfa-2a, RBV 24/48 Week (N=364) | Telaprevir 12 Week+Peg-IFN-alfa-2a, RBV 24/48 Week (N=363)
fatigue (General disorders) | 206 | 211 | 207
influenza like illness (General disorders) | 101 | 105 | 102
pyrexia (General disorders) | 87 | 108 | 95
irritability (General disorders) | 64 | 68 | 80
asthenia (General disorders) | 58 | 62 | 56
chills (General disorders) | 54 | 65 | 46
injection site erythema (General disorders) | 33 | 46 | 38
pain (General disorders) | 28 | 30 | 18
pruritus (Skin and subcutaneous tissue disorders) | 131 | 165 | 181
rash (Skin and subcutaneous tissue disorders) | 88 | 129 | 133
alopecia (Skin and subcutaneous tissue disorders) | 73 | 81 | 83
dry skin (Skin and subcutaneous tissue disorders) | 66 | 66 | 63
rash papular (Skin and subcutaneous tissue disorders) | 15 | 20 | 24
pruritus generalised (Skin and subcutaneous tissue disorders) | 13 | 22 | 22
rash erythematous (Skin and subcutaneous tissue disorders) | 16 | 13 | 17
rash pruritic (Skin and subcutaneous tissue disorders) | 11 | 17 | 16
eczema (Skin and subcutaneous tissue disorders) | 14 | 18 | 10
rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 10 | 23
nausea (Gastrointestinal disorders) | 112 | 146 | 156
diarrhoea (Gastrointestinal disorders) | 80 | 115 | 102
vomiting (Gastrointestinal disorders) | 38 | 55 | 55
haemorrhoids (Gastrointestinal disorders) | 13 | 43 | 43
anorectal discomfort (Gastrointestinal disorders) | 13 | 30 | 46
abdominal pain (Gastrointestinal disorders) | 34 | 28 | 20
dyspepsia (Gastrointestinal disorders) | 23 | 15 | 33
constipation (Gastrointestinal disorders) | 12 | 26 | 27
anal pruritus (Gastrointestinal disorders) | 7 | 25 | 31
headache (Nervous system disorders) | 142 | 156 | 148
dizziness (Nervous system disorders) | 49 | 50 | 57
distrubance in attention (Nervous system disorders) | 33 | 29 | 25
dysgeusia (Nervous system disorders) | 14 | 36 | 34
insomnia (Psychiatric disorders) | 111 | 116 | 117
depression (Psychiatric disorders) | 79 | 61 | 66
anxiety (Psychiatric disorders) | 44 | 33 | 35
affect lability (Psychiatric disorders) | 12 | 5 | 17
anaemia (Blood and lymphatic system disorders) | 70 | 141 | 135
neutropenia (Blood and lymphatic system disorders) | 68 | 62 | 51
cough (Respiratory, thoracic and mediastinal disorders) | 86 | 76 | 61
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 50 | 52 | 47
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 23 | 27 | 26
pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 25 | 28
myalgia (Musculoskeletal and connective tissue disorders) | 77 | 76 | 54
arthralgia (Musculoskeletal and connective tissue disorders) | 68 | 56 | 49
back pain (Musculoskeletal and connective tissue disorders) | 43 | 25 | 28
pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 8 | 19
urinary tract infection (Infections and infestations) | 13 | 22 | 17
upper respiratory tract infection (Infections and infestations) | 18 | 19 | 9
anorexia (Metabolism and nutrition disorders) | 39 | 55 | 53
decreased appetite (Metabolism and nutrition disorders) | 30 | 36 | 36
vision blurred (Eye disorders) | 27 | 26 | 29
weight decreased (Investigations) | 22 | 13 | 24
dry mouth (Gastrointestinal disorders) | 15 | 32 | 33
abdominal pain upper (Gastrointestinal disorders) | 27 | 20 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days